CLINICAL TRIAL: NCT03036761
Title: Interest of Auriculotherapy in Prophylaxis of Migraine and Headache in Patients With Migraines
Acronym: Migauric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/58; 2016-A01534-47 (Other: ANSM)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Headache, Migraine
Keywords: Auriculotherapy
MeSH Terms: conditions — Migraine Disorders | interventions — Auriculotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AUR+: Auriculotherapy (Experimental): Patients benefit from 3 sessions of auriculotherapy at one month intervals.
  Interventions: Procedure: Auriculotherapy
- AUR-: No auriculotherapy (No Intervention): Patients do not benefit from auriculotherapy.

INTERVENTIONS:
Procedure: Auriculotherapy — 3 sessions of auriculotherapy at one month intervals.
  Arms: AUR+: Auriculotherapy

SUMMARY:
The aim of the study is to show that auriculotherapy decreases the number of days with painful episodes of migraine and headache after 3 months of treatment

DETAILED DESCRIPTION:
Prospective, multicenter, controlled and randomized study.

At the inclusion:

* initial assessment of migraine and headache attacks of the last 3 months with the migraine/headache/treatment diary;
* quality of life assessment (MIDAS questionnaire).

Patients are randomized in 2 groups (distribution 2/3 AUR+, 1/3 AUR-):

* AUR+: experimental group "Auriculotherapy". Patients benefit from 3 sessions of auriculotherapy at one month intervals.
* AUR-: control group. Patients do not benefit from auriculotherapy.

After 3 months, a visit of Algology is carried out :

* final assessment of migraine and headache attacks of the last 3 months with the migraine/headache/treatment diary;
* quality of life assessment (MIDAS questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Woman;
* Aged from 18 to 80;
* Benefiting from social security scheme or legal successor;
* Having given their non-opposition to the study; ·
* Diagnosis of chronical migraine for more than 6 months;
* Without background treatment or with stable background therapy for more than 1 month;
* Presenting a calendar of migraines and headaches mentioning the number of days with pain, intensity of pain and treatments for at least 3 months.

Non inclusion Criteria:

* Man;
* Patient with less than 6 painful episodes in 3 months;
* History or actual mental health disorder;
* Dependence on opioids or tranquillizers;
* Secondary headaches;
* Incapacitated to keep a diary of the migraines / headaches / treatments;
* Contraindications for the use of auriculotherapy (scheduled Magnetic resonance imaging examination, declared pregnancy, breastfeeding, artificial heart valves, Haemophilia, effective anticoagulation treatment);
* Having received auriculotherapy treatment in the indication of the study in the last 12 months before inclusion;
* Scheduled to start a new drug or non-drug therapy which could interfere with the study (antidepressant, opioids, anticonvulsant psychological therapy, physiotherapy, deep brain stimulation, etc..);
* Modification of background treatment during the month before inclusion.

Exclusion criteria

* Allergy or infection of the auricle
* Pregnancy

Ages: 18 Months to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 90 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Number of days with migraine and non-migraine headache post inclusion. | 3 months
  Evaluated with the patient's migraine/headache/treatment diary of the last 3 months after inclusion.
  One day with painful episodes of migraines and non-migraines headaches is a day when:
  * the pain episode lasts more than 4 hours,
  * or the pain episode is suppressed by a specific treatment known to the patient.

SECONDARY OUTCOMES:
Number of days with migraine post inclusion. | 3 months
  Evaluated with the patient's migraine/headache/treatment diay of the last 3 months after inclusion.
  One day with painful episodes of migraines is a day when:
  * the pain episode lasts more than 4 hours,
  * or the pain episode is suppressed by a specific treatment known to the patient.
Number of days with non migraine headache post inclusion. | 3 months
  Evaluated with the patient's migraine/headache/treatment diary of the last 3 months after inclusion.
  One day with painful episodes of non-migraines headaches is a day when:
  * the pain episode lasts more than 4 hours,
  * or the pain episode is suppressed by a specific treatment known to the patient.
Intensity of pain episodes (migraines and non-migraine headaches) post inclusion: numerical scale | 3 months
  The intensity of the pain episodes is evaluated by the patient on a numerical scale of 1 to 3 (1 = low, 2 = moderate, 3 = intense) which is in the patient's migraine/headache/treatment diary of the 3 months after inclusion.
  The outcome is evaluated by the calculation of the sum of the pain intensities of migraines and non-migraine headaches .
Evolution of antalgic use (triptan and non-triptan) in migraine patients. | 3 months
  Evaluated with the patient's migraine/headache/treatment diary of the last 3 months after inclusion.
  The sum of antalgic use (triptan and non-triptan):
  * total number of triptan taken;
  * number of days with triptan;
  * total number of non-triptan analgesics taken;
  * number of days with non-triptan analgesics.
Evaluation of the quality of life of the patient: MIDAS score | 3 months
  Calculation of the MIDAS score during the inclusion visit and 3 months after the inclusion visit.
Tolerance of auriculotherapy treatment | 3 months
  The presence or absence of adverse events attributed to the treatment of auriculotherapy by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - Cabinet Médical, Maisons-Alfort
  - Centre Médical de L'Olivier, Montigny-le-Bretonneux
  - GHP Saint Joseph, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Michel-Cherqui M, Ma S, d'Ussel M, Ebbo D, Spassova A, Chaix-Couturier C, Szekely B, Fischler M, Lemaire N, Le Guen M. Auriculotherapy in prevention of migraine attacks: an open randomized trial. Front Neurol. 2023 May 22;14:1193752. doi: 10.3389/fneur.2023.1193752. eCollection 2023. PMID 37284181